CLINICAL TRIAL: NCT03326622
Title: The Role of Moderate Aerobic Exercise as Determined by Cardiopulmonary Exercise Testing in ALS
Brief Title: Exercise and Disease Progression in Amyotrophic Lateral Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Anna Caroline Braga, Investigator, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FCT - SFRH/BD/78413/2011
Record Dates: First submitted 2017-10-21; First posted 2017-10-31 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; aerobic exercise; functional outcome; non-invasive ventilation; oxygen uptake
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Standard of Care; Range of Motion, Articular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate exercise + standard care (Experimental): This group performed a moderate exercise protocol with training zone determined by Cardiopulmonary Exercise testing added to standard care program based on American Academy of Neurology guidelines.
  Interventions: Other: standard care; Other: moderate exercise
- Standard care (Active Comparator): This group performed a standard care program based on American Academy of Neurology guidelines, without exercise intensity control.
  Interventions: Other: standard care

INTERVENTIONS:
Other: standard care — A standard care program based on American Academy of Neurology guidelines (Range Of Motion (ROM) exercises, gait and balance training )at home or another rehabilitation units without intensity control.
  Other Names: Range of Motion; Gait Training; Balance training
Other: moderate exercise — A moderate exercise protocol two times per week in a treadmill in the lower range of the training zone determined by Cardiopulmonary Exercise Testing, monitored by continuous pulse oximetry evaluation.
  Arms: moderate exercise + standard care

SUMMARY:
This study evaluated the influence of a tailored aerobic exercise protocol on the functional outcome in ALS patients. In addition, the investigators compare some CPET variables collected during exercise testing in both groups.

DETAILED DESCRIPTION:
This work aimed to evaluate the effects of a moderate aerobic exercise with controlled intensity determined by Cardiopulmonary Exercise Testing (CPET) and its role on the functional status in ALS patients versus standard care. Additionally, the investigators explored the performance of CPET variables - oxygen uptake (VO2) expressed in L/min, in percentage of predicted or in metabolic equivalents (METs) at peak effort, at anaerobic threshold (AT), the respiratory compensation point (RCP) when achieved, Dioxide Carbon output in L/min (VCO2) and the minute ventilation in L/min (VE) throughout the study.

Assessments:(diagnostic visit - T0), at study entry (T1) and 6 months after (T2) using:

Functional status by Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R), Respiratory function tests (RFT): Forced Vital Capacity predicted (%FVC) and Oxygen saturation provided by pulse oximetry.

CPET was performed in both groups at study entry and 6 months later (T1 and T2), using a treadmill (WOODWAY®) coupled with a gas exchange analyzer (METALYZER® 3B) with ergo-spirometry system using a breath-by-breath technology developed by CORTEX® systems.

Intervention:

G1(Interventional group) performed moderate exercise protocol two times/week in a treadmill in the lower range of the training zone determined by CPET + standard care (range of motion exercise, gait and balance training under continuous pulse oximetry observation).

G2 (control group) performed a standard care exercise program at home or at other rehabilitation units without pulse oximetry observation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients diagnosed with definite, probable, or probable laboratory supported ALS
* Disease duration from first symptoms between 6-24 months to exclude slow and fast progression
* ALSFRS-R ≥ 30
* FVC (%predicted) ≥ 70%

Exclusion Criteria:

* Other medical conditions, like cardiac insufficiency and lung disorders or others conditions limiting exercise training;
* Heavy smoking habits with laboratorial evidence of significant bronchial constriction;
* Signs of associated dementia or psychiatric disorders.

Note: None of the patients were on tube feeding, invasive or non-invasive mechanical ventilation at admission of study protocol (T1).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Functional decline between start and end of the study | between baseline and 6 months later
  It was used the Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R),which rates the functionality of the ALS patients in performing activities involving 4 different areas through 3 sub-scores - bulbar, spinal [upper and lower limb] and also the respiratory function. Each of its questions is rated from 0 (total inability) to 4 points (no functional limitation). The last three questions address the respiratory function (dyspnea, orthopnea, respiratory insufficiency) and assess the respiratory functional outcome.
  The sub-scores rating: Bulbar sub-score between 0 - 12, the spinal score between 0 - 24 and the respiratory sub-score between 0 - 12.The sum of the sub-scores provide an ALSFRS-R total score = 48. Higher values represent a better functionality.

SECONDARY OUTCOMES:
Performance of Cardiopulmonary Exercise testing variables throughout the study | at study entry and 6 months later.
  Changes on the oxygen uptake (VO2peak) measurement following an aerobic exercise protocol compared to standard care.
Changes on the Dioxide Carbon output (VCO2) measurement | at study entry and 6 months later
  Changes on the Dioxide Carbon output (VCO2) following an aerobic exercise protocol compared to standard care.
Changes on the Minute Ventilation (VE) measurement | at study entry and 6 months later
  Changes on Minute ventilation (VE) following an aerobic exercise protocol compared to standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Mamede de Carvalho, MD PhD, Study Director — Institute of Molecular Medicine; Anabela Pinto, MD PhD, Principal Investigator — Institute of Molecular Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization - Physical activity Fact Sheet nº385. In www.who.int/mediacentre/factsheets/fs385/en/ January; 2015
- [Background] Mahoney DJ, Rodriguez C, Devries M, Yasuda N, Tarnopolsky MA. Effects of high-intensity endurance exercise training in the G93A mouse model of amyotrophic lateral sclerosis. Muscle Nerve. 2004 May;29(5):656-62. doi: 10.1002/mus.20004. PMID 15116368
- [Background] Pinto S, Swash M, de Carvalho M. Respiratory exercise in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2012 Jan;13(1):33-43. doi: 10.3109/17482968.2011.626052. PMID 22214352
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Binder RK, Wonisch M, Corra U, Cohen-Solal A, Vanhees L, Saner H, Schmid JP. Methodological approach to the first and second lactate threshold in incremental cardiopulmonary exercise testing. Eur J Cardiovasc Prev Rehabil. 2008 Dec;15(6):726-34. doi: 10.1097/HJR.0b013e328304fed4. PMID 19050438
- [Background] Majmudar S, Wu J, Paganoni S. Rehabilitation in amyotrophic lateral sclerosis: why it matters. Muscle Nerve. 2014 Jul;50(1):4-13. doi: 10.1002/mus.24202. Epub 2014 May 17. PMID 24510737
- [Background] Cup EH, Pieterse AJ, Ten Broek-Pastoor JM, Munneke M, van Engelen BG, Hendricks HT, van der Wilt GJ, Oostendorp RA. Exercise therapy and other types of physical therapy for patients with neuromuscular diseases: a systematic review. Arch Phys Med Rehabil. 2007 Nov;88(11):1452-64. doi: 10.1016/j.apmr.2007.07.024. PMID 17964887
- [Background] Beal MF. Does impairment of energy metabolism result in excitotoxic neuronal death in neurodegenerative illnesses? Ann Neurol. 1992 Feb;31(2):119-30. doi: 10.1002/ana.410310202. PMID 1349466
- [Background] Miller RG, Jackson CE, Kasarskis EJ, England JD, Forshew D, Johnston W, Kalra S, Katz JS, Mitsumoto H, Rosenfeld J, Shoesmith C, Strong MJ, Woolley SC; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter update: the care of the patient with amyotrophic lateral sclerosis: drug, nutritional, and respiratory therapies (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2009 Oct 13;73(15):1218-26. doi: 10.1212/WNL.0b013e3181bc0141. PMID 19822872
- [Background] Pinto AC, Evangelista T, Carvalho M, Alves MA, Sales Luis ML. Respiratory assistance with a non-invasive ventilator (Bipap) in MND/ALS patients: survival rates in a controlled trial. J Neurol Sci. 1995 May;129 Suppl:19-26. doi: 10.1016/0022-510x(95)00052-4. PMID 7595610
- [Background] Bourke SC, Tomlinson M, Williams TL, Bullock RE, Shaw PJ, Gibson GJ. Effects of non-invasive ventilation on survival and quality of life in patients with amyotrophic lateral sclerosis: a randomised controlled trial. Lancet Neurol. 2006 Feb;5(2):140-7. doi: 10.1016/S1474-4422(05)70326-4. PMID 16426990
- [Background] Chetta A, Aiello M, Tzani P, Olivieri D. Assessment and monitoring of ventilatory function and cough efficacy in patients with amyotrophic lateral sclerosis. Monaldi Arch Chest Dis. 2007 Mar;67(1):43-52. doi: 10.4081/monaldi.2007.509. PMID 17564284
- [Background] Motor Neurone Disease: The Use of Non-Invasive Ventilation in the Management of Motor Neurone Disease [Internet]. London: National Institute for Health and Clinical Excellence (NICE); 2010 Jul. Available from http://www.ncbi.nlm.nih.gov/books/NBK65383/ PMID 22171400
- [Background] Cedarbaum JM, Stambler N, Malta E, Fuller C, Hilt D, Thurmond B, Nakanishi A. The ALSFRS-R: a revised ALS functional rating scale that incorporates assessments of respiratory function. BDNF ALS Study Group (Phase III). J Neurol Sci. 1999 Oct 31;169(1-2):13-21. doi: 10.1016/s0022-510x(99)00210-5. PMID 10540002
- [Background] Pinto A, de Carvalho M, Evangelista T, Lopes A, Sales-Luis L. Nocturnal pulse oximetry: a new approach to establish the appropriate time for non-invasive ventilation in ALS patients. Amyotroph Lateral Scler Other Motor Neuron Disord. 2003 Apr;4(1):31-5. doi: 10.1080/14660820310006706. PMID 12745616
- [Background] EFNS Task Force on Diagnosis and Management of Amyotrophic Lateral Sclerosis:; Andersen PM, Abrahams S, Borasio GD, de Carvalho M, Chio A, Van Damme P, Hardiman O, Kollewe K, Morrison KE, Petri S, Pradat PF, Silani V, Tomik B, Wasner M, Weber M. EFNS guidelines on the clinical management of amyotrophic lateral sclerosis (MALS)--revised report of an EFNS task force. Eur J Neurol. 2012 Mar;19(3):360-75. doi: 10.1111/j.1468-1331.2011.03501.x. Epub 2011 Sep 14. PMID 21914052
- [Background] Wasserman K, Hansen JE, Sue DY, Stringer WW, Sietsema KE, Sun X-G, Whipp BJ.Principles of Exercise Testing and Interpretation: Including Pathophysiology and Clinical Applications, 5th edn; eds (2012). Lippincott Williams & Wilkins, Philadelphia, USA.ISBN 978-1-60913-899-8
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Vucic S, Krishnan AV, Kiernan MC. Fatigue and activity dependent changes in axonal excitability in amyotrophic lateral sclerosis. J Neurol Neurosurg Psychiatry. 2007 Nov;78(11):1202-8. doi: 10.1136/jnnp.2006.112078. Epub 2007 Mar 19. PMID 17371901
- [Background] Longstreth WT, Nelson LM, Koepsell TD, van Belle G. Hypotheses to explain the association between vigorous physical activity and amyotrophic lateral sclerosis. Med Hypotheses. 1991 Feb;34(2):144-8. doi: 10.1016/0306-9877(91)90183-y. PMID 2041488
- [Background] Anand A, Thakur K, Gupta PK. ALS and oxidative stress: the neurovascular scenario. Oxid Med Cell Longev. 2013;2013:635831. doi: 10.1155/2013/635831. Epub 2013 Dec 3. PMID 24367722
- [Background] Sanjak M, Paulson D, Sufit R, Reddan W, Beaulieu D, Erickson L, Shug A, Brooks BR. Physiologic and metabolic response to progressive and prolonged exercise in amyotrophic lateral sclerosis. Neurology. 1987 Jul;37(7):1217-20. doi: 10.1212/wnl.37.7.1217. PMID 3601086
- [Background] Mezzani A, Pisano F, Cavalli A, Tommasi MA, Corra U, Colombo S, Grassi B, Marzorati M, Porcelli S, Morandi L, Giannuzzi P. Reduced exercise capacity in early-stage amyotrophic lateral sclerosis: Role of skeletal muscle. Amyotroph Lateral Scler. 2012 Jan;13(1):87-94. doi: 10.3109/17482968.2011.601463. Epub 2011 Aug 11. PMID 21830991
- [Background] Siciliano G, D'Avino C, Del Corona A, Barsacchi R, Kusmic C, Rocchi A, Pastorini E, Murri L. Impaired oxidative metabolism and lipid peroxidation in exercising muscle from ALS patients. Amyotroph Lateral Scler Other Motor Neuron Disord. 2002 Jun;3(2):57-62. doi: 10.1080/146608202760196011. PMID 12215226
- [Background] Battista RA, Foster C, Andrew J, Wright G, Lucia A, Porcari JP. Physiologic responses during indoor cycling. J Strength Cond Res. 2008 Jul;22(4):1236-41. doi: 10.1519/JSC.0b013e318173dbc4. PMID 18545183
- [Background] Hill DW, Rowell AL. Significance of time to exhaustion during exercise at the velocity associated with VO2max. Eur J Appl Physiol Occup Physiol. 1996;72(4):383-6. doi: 10.1007/BF00599701. PMID 8851910
- [Background] Lunetta C, Lizio A, Sansone VA, Cellotto NM, Maestri E, Bettinelli M, Gatti V, Melazzini MG, Meola G, Corbo M. Strictly monitored exercise programs reduce motor deterioration in ALS: preliminary results of a randomized controlled trial. J Neurol. 2016 Jan;263(1):52-60. doi: 10.1007/s00415-015-7924-z. PMID 26477027
- [Background] Blizzard CA, Southam KA, Dawkins E, Lewis KE, King AE, Clark JA, Dickson TC. Identifying the primary site of pathogenesis in amyotrophic lateral sclerosis - vulnerability of lower motor neurons to proximal excitotoxicity. Dis Model Mech. 2015 Mar;8(3):215-24. doi: 10.1242/dmm.018606. PMID 25740331
- [Background] Carilho R, de Carvalho M, Swash M, Pinto S, Pinto A, Costa J. Vascular endothelial growth factor and amyotrophic lateral sclerosis: the interplay with exercise and noninvasive ventilation. Muscle Nerve. 2014 Apr;49(4):545-50. doi: 10.1002/mus.23955. PMID 23868282
- [Background] Takken T, Groen WG, Hulzebos EH, Ernsting CG, van Hasselt PM, Prinsen BH, Helders PJ, Visser G. Exercise stress testing in children with metabolic or neuromuscular disorders. Int J Pediatr. 2010;2010:254829. doi: 10.1155/2010/254829. Epub 2010 Jul 15. PMID 20706686
- [Background] Lanfranconi F, Ferri A, Corna G, Bonazzi R, Lunetta C, Silani V, Riva N, Rigamonti A, Maggiani A, Ferrarese C, Tremolizzo L. Inefficient skeletal muscle oxidative function flanks impaired motor neuron recruitment in Amyotrophic Lateral Sclerosis during exercise. Sci Rep. 2017 Jun 7;7(1):2951. doi: 10.1038/s41598-017-02811-z. PMID 28592858
- [Background] Paganoni S, Cudkowicz M, Berry JD. Outcome measures in amyotrophic lateral sclerosis clinical trials. Clin Investig (Lond). 2014;4(7):605-618. doi: 10.4155/cli.14.52. PMID 28203356
- [Background] Dal Bello-Haas V, Florence JM. Therapeutic exercise for people with amyotrophic lateral sclerosis or motor neuron disease. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD005229. doi: 10.1002/14651858.CD005229.pub3. PMID 23728653
- [Background] Pinto AC, Alves M, Nogueira A, Evangelista T, Carvalho J, Coelho A, de Carvalho M, Sales-Luis ML. Can amyotrophic lateral sclerosis patients with respiratory insufficiency exercise? J Neurol Sci. 1999 Oct 31;169(1-2):69-75. doi: 10.1016/s0022-510x(99)00218-x. PMID 10540010
- [Derived] Braga ACM, Pinto A, Pinto S, de Carvalho M. The Role of Moderate Aerobic Exercise as Determined by Cardiopulmonary Exercise Testing in ALS. Neurol Res Int. 2018 Jan 31;2018:8218697. doi: 10.1155/2018/8218697. eCollection 2018. PMID 29666705